CLINICAL TRIAL: NCT05329948
Title: The Effect of Haptonomy Application on Pregnancy Adjustment and Prenatal Attachment of Fathers
Brief Title: Application of Haptonomy and Pregnancy Adjustment, Paternal Attachment
Acronym: Haptonomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Sibel ÖZTÜRK, Asst. Prof., Ataturk University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Ataturk University SÖZTÜRK0001
Record Dates: First submitted 2022-01-03; First posted 2022-04-15 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Father-Child Relations
Keywords: fetus; midwifery; pregnancy; haptonomy; father

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- haptonomy application (Experimental): The data will be obtained by applying a pre-test to the pregnant women and their spouses included in the experimental group before the application. After the pre-test data are collected, 5 sessions of haptonomy will be applied to the couples in the experimental group. Each session (Breath awareness and diaphragm breathing 5 minutes, Feminine energy attunement and heart-looking energy work 5 minutes, Physical communication with the baby in the womb with touches 10 minutes, meditation from the heart to the uterus 15 minutes, awareness of the environment, closing breath and feedback 5 minutes) It will be 40 minutes. For the effectiveness and continuity between each session, planning will be made for 3 days to 7 days. The final test will be applied 1 week after the hapatonomy application (after 5 sessions are completed).
  Interventions: Other: Haptonomy application
- Control (No Intervention): no application will be made

INTERVENTIONS:
Other: Haptonomy application — Feeling the fetus by touching the mother's womb with meditation
  Arms: haptonomy application

SUMMARY:
The pregnancy process is experienced not only by the mother, but also by the fathers, so it is thought that the application of haptonomy, which is the science of love, communication and feeling together, will confirm the emotional existence of the baby in the prenatal period, and support the attachment of the father and the adaptation of the mothers to pregnancy.

Therefore, this study; It was aimed to evaluate the effect of haptonomy application on prenatal attachment of fathers and compliance with pregnancy and to contribute to the midwifery literature of the results.

DETAILED DESCRIPTION:
In accordance with the literature review, no similar study was found in our country. The reason for the application of haptonomy in pregnancy is the sense of touch, which develops in the first 2 months of pregnancy and is an emotional sense. The pregnancy process is experienced not only by the mother, but also by the fathers, so it is thought that the application of haptonomy, which is the science of love, communication and feeling together, will confirm the emotional existence of the baby in the prenatal period, and support the attachment of the father and the adaptation of the mothers to pregnancy. Therefore, this study; The aim of this study was to evaluate the effect of haptonomy application on prenatal attachment of fathers and adaptation of pregnant women to pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* At least primary school graduate,
* Being at the 24th and 32nd week of pregnancy
* Living with your partner

Exclusion Criteria:

* Having problems with his wife
* Living apart with his wife
* Pregnant women who have completed the 32nd gestational week

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
The Effect of Haptonomy Application Prenatal Attachment of Fathers | one month
  The research is an experimentally planned randomized controlled trial. The sample of the study consists of pregnant women and their spouses (70 experimental group, 70 control group) between the 24th and 32nd weeks.
  Fetal attachment of prospective fathers was evaluated with the intrauterine father attachment scale. Intrauterine Father Attachment consists of 23 items. A minimum score of 23 and a maximum of 92 points is obtained on the scale. Scale has no cutoff point. High scores obtained indicate high level of attachment of father to fetus before birth; low scores mean that the father's level of prenatal attachment to the fetus is low.

SECONDARY OUTCOMES:
The Effect of Haptonomy Application on Pregnancy Adjustment | one month
  Pregnancy compliance of pregnant women was evaluated with the prenatal self-rating scale. The scale is a 4-point Likert-type scale with 79 items and 7 sub-dimensions. A minimum of 79 and a maximum of 316 points can be obtained for the entire scale. Scale has no cutoff point. Low scores indicate high compliance with pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Sibel ÖZTÜRK, Asst.Prof., Study Director — Atatürk University Faculty of Health Sciences Department of Midwifery Yakutiye/Erzurum; Nazlı AKAR, Phd, Principal Investigator — Kafkas University Faculty of Health Sciences Department of Midwifery Merkez/Kars
Locations (1):
- Kars Harakani Devlet Hastanesi, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The principle of "Informed Consent" by informing the pregnant women and their spouses who meet the research criteria and want to support the research, the principle of "Respect for Autonomy" by stating that they are free to participate in the research, the principle of "Confidentiality and Protection of Confidentiality" by stating that the information of the pregnant women and spouses participating in the research will be kept confidential. will be fulfilled.